CLINICAL TRIAL: NCT07220746
Title: Understanding Cognitive-Academic Bidirectionality in Math Learning Disabilities
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Marcia Barnes, Professor, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 240343; 1R01HD115592-01A1 (NIH)
Record Dates: First submitted 2025-10-21; First posted 2025-10-24 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Math Learning Disability
Keywords: math word problem solving; arithmetic; working memory
MeSH Terms: conditions — Dyscalculia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Coordinated Treatment (Experimental): The coordinated treatment group receives standard-of-care math treatment + computerized working memory training, provided contiguously & with coordinated supports for cross-domain transfer.
  Interventions: Behavioral: Coordinated Treatment
- Math Treatment (Active Comparator): The math treatment group receives standard-of-care math treatment + computerized reading instructional activities.
  Interventions: Behavioral: Math Treatment
- Control (No Intervention): The control group receives only the conventional school program, including classroom instruction and school-provided intervention.

INTERVENTIONS:
Behavioral: Coordinated Treatment — Coordinated Treatment provides 15 weeks (3 35-minute sessions per week) of intervention. Each session comprises 2 components delivered contiguously by the same tutor: 15 min of working memory training, immediately followed by 20 min of math (arithmetic & word-problem solving)intervention. Explicit transfer instruction is woven into both components.
  Arms: Coordinated Treatment
Behavioral: Math Treatment — Math Treatment provides 15 weeks (three 35-minute sessions per week) of intervention. Each session comprises 2 components delivered contiguously by the same tutor: 15 min of computerized reading instruction, immediately followed by 20 min of math (arithmetic & word-problem solving) intervention.
  Arms: Math Treatment

SUMMARY:
The goal of this clinical trial is to test the effects of an innovative intervention designed to improve math skills in first graders at risk for math disabilities. The main questions the trial aims to answer are:

* Does combining a math word problem solving intervention with a working memory intervention improve math to a greater extent than the same math intervention without cognitive training?
* Do the findings provide evidence for bidirectional effects on development? In other words, does working memory support math learning and does math learning support working memory development?

Screening for eligibility will take place in two testing sessions. Students who meet the eligibility criteria will be randomly assigned to one of three groups:

1. One treatment group will receive a validated treatment for math word problem solving plus computerized working memory training.
2. Another treatment group will receive the same validated math treatment plus computerized reading instruction.
3. A control group will receive the conventional school math program, including any additional school-provided intervention.

Participants in both treatment groups will receive 35 minutes of tutoring three times per week for 15 weeks.

Children who are selected to participate in the study will be tested once before this project's intervention begins; twice after intervention starts; twice after intervention ends; and once near the end of second grade to see how long effects last.

DETAILED DESCRIPTION:
The focus of this clinical trial (CT) is an innovative intervention guided by cognitive-academic mutualism theory in which cognitive resources support development of academic competencies while academic learning in turn exercises and strengthens cognitive abilities. The goal of this CT is to test the effects of an innovative intervention designed to improve cognitive ability and academic skill in coordinated fashion and test bidirectionality as a mechanistic process by which effects occur, thereby evaluating the potential for cognitive-academic mutualism to expand the framework for learning disabilities intervention science and advancing understanding about the development of mathematic competence in children. The CT's innovative intervention provides coordinated cognitive training + direct skills math intervention, with supports for cross-domain transfer. The academic focus is math: word-problem solving (WPS) & arithmetic, both critical foundational skills. The cognitive focus is complex working memory span (WM) because WM plays a central role in early math development. Participants are 6-8 years old, a sensitive period when WM malleability and beneficial effects between emerging skills are rich in opportunity & when school instruction on the targeted math competencies intensifies.

Participants are 300 children who begin 1st grade with math delays & low WM. They are identified as meeting inclusion criteria using a 2-stage screening process. Children who enter the study complete pretesting & then are randomly assigned to 3 conditions: (1) CO-Tx, standard-of-care math treatment + computerized WM training, provided contiguously & with coordinated supports for cross-domain transfer (the innovation); (2) M-Tx, the same standard-of- care math treatment + the same amount of computerized reading instructional activities (the contrast standard-of-care condition); & (3) CON, the control group (maturation and the conventional school program, including classroom instruction and school-provided intervention). Children in conditions 1 & 2 receive researcher-delivered intervention at their school for 15 weeks (3 times per week, 35-min per session). WM & math are assessed at pretest, 5 weeks later, another 5 weeks later, posttest, delayed posttest, and follow-up. The study is conducted in 5 cohorts, with 1/5 of the sample entering the study each year.

The Overall Goal is to test CO-Tx's added value over standard-of-care (SOC) math intervention (and over conventional school programming & maturation) while deepening understanding of bidirectional influences between WM & math as a mechanism by which CO-Tx's effects occur and providing insight into cognitive-academic mutualism in children with math delays at start of 1st grade. Aim 1 tests CO-Tx's added value over M-Tx (SOC math intervention + computerized reading activities in each session's 1st component to control for CO-Tx's WM training time) and over CON (the control group) on WM and math (Arith & WPS) at posttest & delayed posttest. One-year follow-up effects are explored. Aim 2 assesses (a) whether bidirectional relations between WM & math are involved in the mediation pathway linking CO-Tx's effects on delayed posttest math & WM and (b) whether bidirectional relations are stronger in CO-Tx than other conditions. Exploratory Aim 3 (subgroup effects) provides insight into the robustness of CO-Tx's effects for boys vs. girls, as a function of economic disadvantage, and for native-Spanish-speaking English learners (i.e., who receive English language services) vs. non-English learners (i.e., native English speakers and non-native-English speakers who do not receive English language services), and ADHD symptom level.

This CT impacts science by deepening understanding about the potential of innovative treatment based on cognitive academic mutualism theory to enhance learning over conventional SOC math intervention; by providing insights into cognitive-academic mutualism as a framework for expanding LD intervention science; and more generally by advancing understanding about cognitive-academic mutualism in developmental science. Results may impact clinical practice by providing proof-of-concept evidence on an innovative approach for advancing LD intervention science. This CT is relevant significant & relevant because math disabilities are associated with poor school, employment, everyday life, & mental health outcomes and given the pressing need to expand the framework for treating LDs.

ELIGIBILITY:
Inclusion Criteria:

* Attends a participating school in the Metropolitan-Nashville Public Schools
* Is a member of a first-grade classroom whose teacher has agreed to let his/her students participate
* Has the available school schedule to participate
* Scores below the 30th percentile on the study's screening math test
* Scores below the 50th percentile on the study's working memory test
* Scores at or above the 7th percentile on at least one of the study's two measures of cognitive performance

Exclusion Criterion:

* Does not attend a participating school in the Metropolitan-Nashville Public Schools
* Is not a member of a first-grade classroom whose teacher has agreed to let his/her students participate
* Does not have the available school schedule to participate
* Scores at or above 30th percentile on the study's screening math test
* Scores at or above the 50th percentile on the study's screening working test
* Scores below the 7th percentile on both of the study's two measures of cognitive performance

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2030-04-30 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Arithmetic Combinations (Fuchs et al., 2003) | Pretest before treatment begins, 5 weeks after treatment starts, 10 weeks after treatment starts, 15 weeks after treatment starts, 20 weeks after treatment starts, 1 year + 20 weeks after treatment starts
  Children have 1 minute to write answers to 25 addition items (sums 5-12); 1 minute same for subtraction items (minuends 5-12); same 1 minute for 25 addition items (sums 5-18); same and 1 minute for 25 subtraction items (minuends 5-18).
Pennies Story Problems (Jordan & Hanich, 2000) (Jordan & Hanich, 2000) | Pretest before treatment begins, 5 weeks after treatment starts, 10 weeks after treatment starts, 15 weeks after treatment starts
  The test comprises 14 combine, compare and change word problems, each involving penny scenarios and requiring sums and minuends to 12. Items are scored for correct math.
Word Problem Test (Fuchs et al., 2021) | Pretest before treatment begins, 5 weeks after treatment starts, 10 weeks after treatment starts, 15 weeks after treatment starts, 20 weeks after treatment starts, 1 year + 20 weeks after treatment starts
  The test comprises 12 combine, compare and change word problems, some with irrelevant information and/or transfer features (e.g., relevant numbers in graphs and tables, implicit change verbs (e.g. Lost). Items are scored for correct arithmetic and correct label to reflect understanding of both the word problem narrative (i.e,, that the child includes the label "trucks" in their answer if the story had to do with transforming quantitative information having to do with the number of trucks), and the mathematics required to accurately solve the problem.
Working Memory Assessment-Odd-One Out (Alloway, 2012) | Pretest before treatment begins, 5 weeks after treatment starts, 10 weeks after treatment starts, 15 weeks after treatment starts, 20 weeks after treatment starts, 1 year + 20 weeks after treatment starts
  Children see 3 shapes, each in a box shown in a row, and identify the odd-one-out; after making odd-one-out determinations for a series of rows, they recall the location of each odd-one-out shape in order by tapping boxes.
Working Memory Test Battery - Children - Listening Recall (Pickering & Gathercole, 2001) | Pretest before treatment begins, 5 weeks after treatment starts, 10 weeks after treatment starts, 15 weeks after treatment starts, 20 weeks after treatment starts, 1 year + 20 weeks after treatment starts
  Children decide if a sentence is true; after making true/false determinations for a series of sentences, they recall the last word of each sentence in order.
Working Memory Test Battery- Children - Counting Recall (Pickering & Gathercole, 2001) | Pretest before treatment begins, 5 weeks after treatment starts, 10 weeks after treatment starts, 15 weeks after treatment starts, 20 weeks after treatment starts, 1 year + 20 weeks after treatment starts
  Children count a set of 4, 5, 6, or 7 dots on a card; after counting a series of cards, they recall the counts in order.
Wide Range Achievement Test-5-Math | Pretest before treatment begins, 15 weeks after treatment starts, 1 year + 20 weeks after treatment starts
  Test includes an oral section on early numerical competencies (e.g., counting) & a 10-min written section on calculations.
GMADE-Problem Solving & Procedures | 15 weeks after treatment starts, 1 year + 20 weeks after treatment starts
  Tests assesses word problem solving and math applications with 28 items.

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Research staff will make de-identified data sets electronically available to external users under a data-sharing agreement providing the user's commitment to use data for the research purposes described in the user's request; assurance that no research participant will be identified for any purpose; a commitment to securing the data; a commitment to not transferring data to other users & destroying the data after analyses are complete; & guarantees publications are credited to grant/agency and entered in PubMed. Once the user signs and returns the Agreement Form, a database with the variables of interest and codebook are provided, and staff provide relevant, de-identified data and segments of the code book with variable names/values, notes clarifying scoring/data-reduction methods not otherwise available, and a technical report describing the sample, study, and procedures.
Supporting Information: Study Protocol, SAP
Time Frame: The de-identified (stripped) primary outcome data set will become available no later than acceptance for publication of the main findings from the final data set and remain accessible for 3 years following the closeout of this grant. This time frame for data accessibility will be reviewed at the proposed project's completion and revised as needed.
  If all Investigators leave or become unavailable, the last remaining Investigator will assume responsibility for identifying a Vanderbilt faculty member to undertake these responsibilities.
Access Criteria: The user submits a request describing variables of interest, research aims, & quantitative methods and signs a user agreement form (see Plan Description).
URL: https://ldbase.org/